CLINICAL TRIAL: NCT05759195
Title: Tumor Biomolecular Analysis for Defining Predictive Factors for Response to Regorafenib in Recurrent Glioblastoma
Brief Title: Biomolecular Analysis for Predicting Response to Regorafenib
Acronym: RegoRec
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 3458
Record Dates: First submitted 2023-02-23; First posted 2023-03-08 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Glioblastoma; Glioblastoma, IDH-wildtype
Keywords: regorafenib; NGS; predictive biomarker
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biomolecular tumor analysis (Other): NGS, IHC, methylome and other molecular studies
  Interventions: Diagnostic Test: Biomolecular tumor analysis

INTERVENTIONS:
Diagnostic Test: Biomolecular tumor analysis — NGS analysis, other molecular analyses on FFPE tumor tissue

SUMMARY:
The study envisages NGS analysis on tumor tissue from patients treated with regorafenib for recurrent glioblastoma as per standard care, with the aim to identify predictive biomarkers for response.

ELIGIBILITY:
Inclusion Criteria:

1. recurrent glioblastoma after surgery and chemoradiation with temozolomide;
2. indication to treatment with regorafenib per standard of care;
3. written informed consent.

Exclusion Criteria:

None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | through study completion, an average of 3 years
  Interval between tumor diagnosis and death or end of follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No